CLINICAL TRIAL: NCT02343237
Title: A Multicenter, Randomized Study, Against Credible Factitious Intervention That Evaluates the Interest of Osteopathic Medicine in the Management of Fibromyalgia Syndrome
Brief Title: Osteopathic Medicine in Fibromyalgia Syndrome
Acronym: FIBROPATHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130605
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia syndrome; pain; quality of life; osteopathic treatment
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathy + (Experimental): 75 patients will make 6 osteopathic sessions
  Interventions: Procedure: Osteopathic treatment
- Osteopathy - (Active Comparator): 75 patients will make 6 factitious osteopathic sessions
  Interventions: Procedure: Factitious osteopathic treatment

INTERVENTIONS:
Procedure: Osteopathic treatment — osteopathic sessions of 20 minutes
  Arms: Osteopathy +
Procedure: Factitious osteopathic treatment — 6 factitious osteopathic sessions of 20 minutes
  Arms: Osteopathy -

SUMMARY:
The purpose of this study is to evaluate the analgesic effects of a 6 weeks osteopathic treatment on patients with fibromyalgia.

DETAILED DESCRIPTION:
An osteopathic treatment could have a positive and durable effect on pain and quality of life on patients with fibromyalgia.

This technique, in addition to the standard treatment in a multidisciplinary care center, could be efficient by releasing muscle tension.

This is a 24 months multicenter (2 recruiting centers, 1 care center), randomized, and placebo-controlled study. The purpose is to evaluate the analgesic efficacy of a 6 weeks osteopathic treatment compared to a 6 week standard treatment on patients with fibromyalgia. It includes 6 osteopathic/standard sessions of 20 minutes (of one week apart), a follow-up at 3 months, 6 months and 12 months.

The primary aim of this study is to evaluate the pain after each osteopathic session, at the end of the 6 weeks treatment, and after each visit, judging by the patient's pain measured by a numeric scale (EVA).

The secondary aims of this study, based on clinical exams and questionnaires are to evaluate the quality of life, the patient activity and the sleep improvement after osteopathic treatment, and to investigate if osteopathic medicine improves fatigue, comorbidities, and decrease additional visits and medical investigations.

This study will also allow to identify the profile of the osteopathic treatment responders patients

ELIGIBILITY:
Inclusion Criteria:

1. Patient Male or female aged at least of 18
2. Patient with fibromyalgia, according to the American College of Rheumatology (ACR) 1990 criteria, with a global level of pain of 50 over a 100 mm EVA scale
3. Patient suffering from fibromyalgia for over a year
4. Patient with stable medical/non medical treatment for at least 1 month before the recruitment
5. Patient referred to a medical center for a multidisciplinary approach
6. Patient who can be followed for at least 12 months after the end of the osteopathic sessions
7. Patient giving his informed consent to participate in the study
8. Patient affiliated to or beneficiary of social insurance

Exclusion Criteria:

1. Treatment by physical approach in progress or not older than 3 months : physiotherapy, kinesitherapy, rehabilitation or manual treatment (osteopathic or chiropractic care, manual medicine)
2. Unability to attend 6 sessions, meaning one weekly session, of osteopathy, at Hôtel Dieu
3. Severe psychiatric pathology : major depression, psychosis
4. Pregnancy or breast feeding
5. The patient is already included in another clinical study
6. Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain during the 6 weeks of osteopathic treatment | 6 weeks
  The assessment will be on the declarative of the patient. He will report every week the intensity of pain measured by a numeric scale (0 to 100).

SECONDARY OUTCOMES:
Quality of life | 6 weeks after osteopathic treatment
  Questionnaires: Fibromyalgia Impact Questionnaire (FIQ) and SF-36 (Short Form health survey)
Quality of life | 3 months after osteopathic treatment
  Questionnaires: FIQ and SF-36
Quality of life | 6 months after osteopathic treatment
  Questionnaires: FIQ and SF-36
Quality of life | 1 year after osteopathic treatment
  Questionnaires: FIQ and SF-36
Fatigue | 6 weeks after osteopathic treatment
  Questionnaires: multidimensional fatigue inventory (MFI) scale
Fatigue | 3 months after osteopathic treatment
  Questionnaires: MFI scale
Fatigue | 6 months after osteopathic treatment
  Questionnaires: MFI scale
Fatigue | 1 year after osteopathic treatment
  Questionnaires: MFI scale
Pain | 6 weeks after osteopathic treatment
  Questionnaires: Brief Pain Inventory (BPI)
Pain | 3 months after osteopathic treatment
  Questionnaires: BPI
Pain | 6 months after osteopathic treatment
  Questionnaires: BPI
Pain | 1 year after osteopathic treatment
  Questionnaires: BPI

CONTACTS AND LOCATIONS:
Overall Officials: Serge PERROT, PU-PH, Principal Investigator — + 33 1.42.34.84.49
Locations (1):
- Hotel-Dieu Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coste J, Medkour T, Maigne JY, Perez M, Laroche F, Perrot S. Osteopathic medicine for fibromyalgia: a sham-controlled randomized clinical trial. Ther Adv Musculoskelet Dis. 2021 Apr 16;13:1759720X211009017. doi: 10.1177/1759720X211009017. eCollection 2021. PMID 33948127